CLINICAL TRIAL: NCT07108244
Title: Use of [18F]FET PET-MRI to Improve Detection of Pituitary Adenomas in Cushing's Disease - a Prospective Diagnostic Study
Brief Title: Use of [18F]FET PET-MRI to Improve Detection of Pituitary Adenomas in Cushing's Disease
Acronym: FIND
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Erasmus Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FIND study
Record Dates: First submitted 2025-07-25; First posted 2025-08-06 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Cushing Disease
MeSH Terms: conditions — Pituitary ACTH Hypersecretion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [18F]FET-PET-MRI vs IPSS for diagnosing CD vs ectopic CS in ACTH-dependent cases (Other): Participants will undergo both [18F]FET-PET-MRI and inferior petrosal sinus sampling (IPSS) to evaluate their diagnostic performance in differentiating Cushing's disease from ectopic ACTH secretion. Results of both procedures will be made available to the treating medical team and participants as they become available.
  Interventions: Diagnostic Test: [18F]FET PET-MRI

INTERVENTIONS:
Diagnostic Test: [18F]FET PET-MRI — All participants will undergo both [18F]fluoroethyltyrosine positron emission tomography-magnetic resonance imaging ([18F]FET-PET-MRI) and inferior petrosal sinus sampling (IPSS) as part of the diagnostic work-up for ACTH-dependent hypercortisolism. The purpose is to compare the diagnostic accuracy of these two modalities in distinguishing Cushing's disease from ectopic ACTH secretion. The results from both diagnostic tests will be communicated to the treating medical team and the participant to guide further clinical management.

SUMMARY:
In ACTH-dependent hypercortisolism it is important to distinguish between Cushing's disease (CD), with ACTH production by a pituitary neuroendocrine tumour (PitNET) and Cushing's syndrome (CS), with ectopic ACTH production. Bilateral inferior petrosal sinus sampling (IPSS) is the gold standard for this distinction, with a diagnostic accuracy of 98%. However, IPSS is an invasive procedure and an indi-rect diagnostic method, rarely providing reliable data on the exact location of the PitNET. This has a major impact on the therapeutic approach, short and long-term remission rates, and other outcomes. Hybrid Positron-emission tomography-Magnetic Resonance Imaging (PET-MRI) using O-(2-[18F]-fluo-roethyl)-L-tyrosine ([18F]FET) is promising in this respect. Recent data published by our research group demonstrate a a sensitivity of 100% a high accuracy in in the precise localization of ACTH-secreting PitNETs. We hypothesize that [18F]FET PET-MRI could become the new non-invasive diagnostic stand-ard, but data regarding a direct comparison between the diagnostic impact of [18F]FET PET-MRI versus IPSS in the differentiation between CD and ectopic CS are lacking. In addition, there are currently no other reliable biomarkers to distinguish the two disorders. The investigators hypothesize that the ACTH-dependent biomarker copeptin could be a valuable addition in this regard. The aim of this prospective diagnostic study is to compare the diagnostic accuracy of [18F]FET-PET-MRI and IPSS in differentiating CD from ectopic CS in patients with ACTH-dependent hypercortisolism.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Biochemically confirmed ACTH-dependent hypercortisolism, defined as:
* Non-suppressed ACTH levels plus minimal 2 of the following:
* Overnight 1mg dexamethasone suppression test > 50 nmol/L
* Elevated late night salivary cortisol (min. 2/3 measurements)
* Elevated 24-hours urinary free cortisol (min. 2 measurements)
* Pituitary microadenoma (< 10mm) OR negative / inconclusive findings on standard MRI of the pituitary sella-region.
* Indication for further evaluation with IPSS

Exclusion Criteria:

* Non-ACTH dependent hypercortisolism
* Pituitary macroadenoma (≥ 10mm)
* Suspicion of Pseudo-Cushing's disease (e.g. due to alcohol use disorder, PCO's, obesity, de-pression) according to standard work up / guidelines
* use of glucocorticosteroids
* Impaired renal function, defined as eGFR (MDRD) <30ml/min/1,73 m2. An exception can be made in consultation with the treating physician.
* Impaired Liver function
* Pregnancy/breastfeeding. For the latter, temporary discontinuation may be considered.
* Known allergic reaction to therapeutic radiopharmaceuticals.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2025-10-22 (Actual); Primary Completion 2029-07-30 (Estimated); Study Completion 2029-07-30 (Estimated)

PRIMARY OUTCOMES:
Comparison of the proportion of correct distinctions between CD and ectopic CS in patients with ACTH-dependent hypercortisolism using [18F]FET PET-MRI versus IPSS | Patients will receive standard surgical or radiotherapeutic treatment. The study will collect follow-up data 3-6 months post-treatment without influencing clinical management or requiring study-specific visits.
  The difference in the proportion of correct distinction between CD and ectopic CS in patients with ACTH-dependent hypercortisolism using [18F]FET PET-MRI versus IPSS

SECONDARY OUTCOMES:
Copeptin values during IPSS | During the IPSS
  Best fit of diagnostic copeptin values for differentiation between CD and ectopic CS with the inferior petrosal sinus sampling (IPSS) after desmopressin injection,
ACTH values during IPSS | During the IPSS
  Best fit of diagnostic ACTH values for differentiation between CD and ectopic CS with the inferior petrosal sinus sampling (IPSS) after desmopressin injection
Comparison of the diagnostic accuracy between [18F]FET PET-MRI and IPSS for differentiating between CD and ectopic CS in patients with ACTH-dependent hy-percortisolism | Follow-up data 3-6 months post-treatment
  ROC AUC of the [18F]FET PET-MRI and IPSS in differentiating CD from ectopic CS Sensitivity, specificity, positive predictive value (PPV) and negative predictive value (NPV) of the [18F]FET PET-MRI and IPSS for differentiation between CD and ectopic CS
Exact localization of small functional PitNETs in patients with CD using the [18F]FET PET-MRI | perioperative
  Stated as left, central or right side, assessed by an experienced nuclear medicine physician and neuroradiologist Sensitivity, specificity, PPV and NPV of the [18F]FET PET-MRI for the exact localization of small functional PitNETs in patients with CD
Exact localization of small functional PitNETs in patients with CD using the inferior petrosal sinus sampling (IPSS) | perioperative
  Sensitivity, specificity, PPV and NPV of the IPSS for the exact localization of small functional PitNETs in patients with CD
Exact localization of small functional PitNETs in patients with CD using the structural MRI | perioperative
  Sensitivity, specificity, PPV and NPV of the structural MRI for the exact localization of small functional PitNETs in patients with CD

CONTACTS AND LOCATIONS:
Locations (2):
- Erasmus University Medical Centre, Rotterdam, South Holland, Netherlands
- University Hospital Basel, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: No